CLINICAL TRIAL: NCT05074615
Title: Effects of Cranio-cervical Flexion Training on Cervical Proprioception in Patients With Mechanical Neck Pain
Brief Title: Effects of Cranio-cervical Flexion on Cervical Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00945 Laiba Gul
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Neck Pain
Keywords: Mechanical neck pain; Proprioceptive training; Deep cervical flexors
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranio-Cervical Flexion Training Group (Experimental): Participants of this group will receive conventional training along with cranio-cervical flexion training and home plan.
  Cranio-cervical flexion training will be given with the help of pressure biofeedback unit. the cuff will be inflated at a specific pressure level and patient will be asked to maintain that pressure and gradually increase it.
  Interventions: Other: Cranio-Cervical Flexion Training; Other: Conventional Therapy
- Conventional Therapy Group (Active Comparator): Participants of this group will receive only conventional therapy and home plan will be given which includes; hot pack, TENS, neck isometrics and passive stretching of neck musculature. Home plan will include self-stretches and neck isometrics.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Cranio-Cervical Flexion Training — Participants of this group will receive conventional training along with Cranio-cervical flexion training:
  * The pressure cuff is placed behind the neck just next to the occiput and inflated up to a baseline pressure of 20 mmHg. The patient is asked to perform Cranio-Cervical Flexion (CCF) to sequentially reach 5 pressure targets in 2 mmHg increments from a baseline of 20 mmHg to the final level of 30 mmHg. For each target level, the patient is instructed to maintain the contraction for 10 sec for 10 repetitions with brief rest periods between each contraction i.e., 3-5 seconds. Once a set of 10 repetitions of 10 sec is achieved at one target level, the exercise is progressed to train at the next target level up to the final target level at 30 mmHg.
  Conventional therapy will be given along with home plan. Exercise protocol will consist of 30 minutes. Exercise will have total 3 sessions/week for 3 weeks.
  Arms: Cranio-Cervical Flexion Training Group
Other: Conventional Therapy — Participants of this group will receive only conventional therapy and home plan will be given which includes;
  * Hot pack placed on the posterior neck for 15 minutes.
  * Transcutaneous electrical nerve stimulation (TENS) with a frequency of 80 Hz for 20 minutes with 10-30 mA intensity.
  * Isometric exercises: Isometric neck flexion, extension, side bending exercises. 10 repetitions. Hold period is 10 seconds for each movement. Resistance would be provided manually by the therapist.
  * Stretching exercises: Passive stretching for Sternocleidomastoid, Trapezius, Pectoralis Major. 10 reps and each stretch maintained for 10 seconds.
  * Home Plan: Patients will be given a home plan of self-stretches and isometrics and instructions on how to perform and number of repetitions will be guided. Exercise protocol will consist of 25 minutes. Exercise will consist of total 3 sessions/week for 3 weeks

SUMMARY:
To determine the effects of cranio-cervical flexion training on the cervical proprioception and pain in patients with mechanical neck pain.

DETAILED DESCRIPTION:
Neck pain is a very common health related problem that alters an individual's daily life. In the over-all population and musculoskeletal training, it happens next to low back pain in its frequency. Neck pain has a point incidence of approximately 13% and a lifetime incidence of almost 50%. It is a joint reason for visits in accidents and emergency departments. Neck pain is said to be more common in females than in males and it crests at the middle age. Sedentary lifestyles are contributing to the occurrence of neck pain. Chronic neck pain affects a very significant number when it comes to the adult population. Proprioception involves the body sensations that helps in the proper orientation of the body relative to the movement of joints and bones, in rest and in motion. When the joint position sense is disturbed due to some kind of abnormality, a person adopts an abnormal posture. If this faulty posture continues, this causes abnormalities in the spine and causes impaired stability. The system of proprioception in our body is dependent upon different afferent stimulus reaching towards mechanoreceptors from afferent neurons. Due to the presence of high densities of muscle spindles in the slow twitch fibers in deep, small intrinsic dorsal and sub-occipital muscles play very important role in the control of posture. The cervical musculature has a number of other systems working in congregation including vestibular system, visual as well as central nervous system feedbacks. All of these systems send the signals according to the body and head movements. That is why, the involvement of upper cervical region can cause impaired proprioception and altered afferent stimulus. When many levels of nervous system gets involved, it can impact a change in the sensitivity of muscle spindle and causes one of the major proprioception shortages in cervical patients. For the maintenance of motion, posture and joint position, proprioceptive information has an important role and any factor that disrupts this information may be considered a major reason of incorrect motion patterns and symptoms of chronic recurrent pain.

Cranio-Cervical flexion training which aims to enhance activation of the Deep Cervical flexors (DCFs) and restore coordination between the deep and superficial cervical flexors, is one form of exercise that has been advocated for addressing impaired neuromuscular control of the cervical flexors. Clinical trials examining the effectiveness of this exercise regime have demonstrated positive outcomes in terms of decrease in neck pain and disability, improvement in sitting posture, enhanced neuromuscular control of the cervical flexors in patients with chronic neck pain and also improved proprioceptive acuity of the neck, indicating that proprioception can be enhanced with specific exercise. Cranio-cervical flexion training will be done using Pressure Biofeedback Device by Chattanooga.

A cervical range of motion (CROM) device will be used to assess cervical proprioception. The unit of CROM has three inclinometers attached to it and each inclinometer collects degree of movement in each plane. The CROM device has an advantage over the use of a single inclinometer that it does not have to be moved again to measure the degree of movements in other planes. One the CROM device is mounted on the patient's head, instructions are given to the patient regarding their neutral head movements and target head movements. After that, patient is blindfolded and all the movements are performed with patient being blindfolded. No feedback should be given during the ongoing session. This entire procedure takes around 15 minutes for one individual.

In the light of previous research works, the disturbances in the proprioception involving cervical spine are a very important factor in treating the patients with neck pains. It is very important for a physical therapist to address these deficits and stop the vicious cycle of pain as well as improve proprioception. So, this study is aimed at improving the proprioception and decreasing mechanical neck pain with the help of deep cervical muscles flexion training using pressure biofeedback device.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mechanical neck pain with minimum duration of 4 weeks,
* Pain in the cervical region with moving or palpating the cervical spine,
* upper cervical involvement with or without headache and C1-C2 rotational deficits.

Exclusion Criteria:

* Vertebrobasilar insufficiency.
* Any history of serious underlying pathology, cervical trauma, structural deformities, genetic spinal disorders or previous spinal surgery.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Cervical Range of Motion | 3 weeks
  The unit of CROM has three inclinometers attached to it and each inclinometer collects degree of movement in each plane.. One the CROM device is mounted on the patient's head, instructions are given to the patient regarding their neutral head movements and target head movements which are Right and Left sided rotation, Right and Left sided lateral flexion and cervical flexion and extension. After that, patient is blindfolded and all the movements are performed with patient being blindfolded. No feedback should be given during the ongoing session. This entire procedure takes around 15 minutes for one individual.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 3 weeks
  Numeric Pain Rating Scale will be used to measure the level of pain of patients. patient will be asked to rate their perceived level of pain from 0 to 10. 0 being no pain and 10 means highest.

CONTACTS AND LOCATIONS:
Overall Officials: Saad Rauf, Master, Principal Investigator — Riphah International University
Locations (1):
- SPIRE Medical Mall, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No